CLINICAL TRIAL: NCT04752449
Title: Virtual Cognitive Behavioural Therapy for Psychosis: A Randomized Controlled Trial
Brief Title: Virtual Cognitive Behavioural Therapy for Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Michael Best, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39916
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: cbt; psychosis; schizophrenia; cbtp; cognitive behavioural therapy; psychotherapy; virtual
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either Virtual Cognitive Behavioural Therapy or to Treatment as Usual. All participants who receive Treatment as Usual will be offered CBT at the end of the study period.
Who Masked: Outcomes Assessor
Masking Description: Participants will be informed after their first assessment whether they were randomized to CBTp or TAU. Those in TAU are offered CBTp at the end of the study period. Assessors remain blind throughout the study and therefore do not partake in the treatment intervention. Due to the nature of the study, the treatment providers cannot be blinded as those they treat have clearly been randomized to the CBTp condition. The investigator is not blind to any of the randomization outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Cognitive Behavioural Therapy for Psychosis (Experimental): CBT will be delivered according to an established manual that the PI has previously used successfully for in-person treatment. Treatment will consist of individual sessions with a psychologist employed by the University of Toronto for 1-hour per week for 6-months, or by one of the listed clinical graduate students under his supervision. All treatment will be delivered virtually in the participant's home using the online platform Zoom which is PHIPA/PIPEDA compliant. If participants do not have the technology required for virtual sessions, then a tablet will be loaned to them for the duration of treatment. This treatment will be delivered in addition to usual care and no changes to usual care will be required.
  Interventions: Behavioral: Virtual Cognitive Behavioural Therapy for Psychosis
- Treatment as Usual (No Intervention): Participants continue with their regular standard of care without the addition of virtual Cognitive Behavioural Therapy for Psychosis.

INTERVENTIONS:
Behavioral: Virtual Cognitive Behavioural Therapy for Psychosis — CBT will be delivered according to an established manual that the PI has previously used successfully for in-person treatment. Treatment will consist of individual sessions with a psychologist employed by the University of Toronto for 1-hour per week for 6-months, or by one of the listed clinical graduate students under his supervision. All treatment will be delivered virtually in the participant's home using the online platform Zoom which is PHIPA/PIPEDA compliant. If participants do not have the technology required for virtual sessions, then a tablet will be loaned to them for the duration of treatment. This treatment will be delivered in addition to usual care and no changes to usual care will be required.
  Other Names: CBT; CBTp
  Arms: Virtual Cognitive Behavioural Therapy for Psychosis

SUMMARY:
Participants with schizophrenia-spectrum disorders who are experiencing active symptoms of psychosis will randomized to either receive 6 months of individual cognitive behavioural therapy for psychosis or to receive treatment as usual. Participants will be assessed at baseline, 6 months, and 12 months.

DETAILED DESCRIPTION:
Schizophrenia-spectrum disorders are the most persistent, debilitating, and economically burdensome mental illnesses worldwide, and are associated with the greatest per-patient expense of all mental health conditions. Schizophrenia is associated with a 15-20 year decrease in life expectancy, 5-fold increase in likelihood of death by suicide, and a significant decrease in quality of life. Antipsychotic medications are the first line treatment for individuals with schizophrenia spectrum disorders and are prescribed to nearly every service-user. However, in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) trial (one of the largest antipsychotic trials in 1493 individuals with schizophrenia), medication effects on psychosocial functioning were small (d = 0.25). Thus, the primary treatment available to all individuals with schizophrenia does little to improve community functioning. This may partially be a result of the limited efficacy of antipsychotic medication to improve neurocognitive abilities, widely recognized as a core feature of schizophrenia, and one recommendation stemming from the CATIE trial was that "more intensive psychosocial rehabilitative services, including cognitive rehabilitation, may be needed to affect more substantial gains in functioning."

Cognitive behavioural therapy (CBT) is a psychological intervention originally developed to treat depression, and subsequently adapted to treat schizophrenia spectrum disorders. CBT has demonstrated moderate treatment effects (d = 0.36 - 0.44) in multiple meta-analyses and is widely recommended for the treatment of schizophrenia in international guidelines. CBT involves clients learning to evaluate their cognitive content in order to develop more accurate representations of the world. CBT has proven effective for improving hallucinations, delusions, negative symptoms, and personal recovery.

Despite the established efficacy of CBT delivered through in-person methods, most clinics have discontinued in-person treatments as a result of the COVID-19 pandemic and have moved to virtual delivery methods. While it has been assumed that virtual delivery of CBT is equivalent to in-person delivery, our recent systematic review demonstrated that there has never been a trial examining the efficacy of virtually delivered CBT for psychosis. Characteristics of schizophrenia such as paranoia, and disorganization already present challenges to psychological treatment and it is possible that this challenge will be further exacerbated by treatment delivery through virtual methods. Additionally, it is unclear the extent to which individuals with schizophrenia-spectrum disorders will be interested in receiving virtual CBT and capable of using the technology that is required.

Thus the goals of the current study are two-fold:

1. Examine the efficacy of virtually delivered CBT for schizophrenia-spectrum disorders to reduce symptoms and improve community functioning.
2. Examine the feasibility and acceptability of virtually-delivered CBT for individuals with schizophrenia-spectrum disorders.

CBT will be delivered according to an established manual that the PI has previously used successfully for in-person treatment. Treatment will consist of individual sessions with a therapist for 1-hour per week for 6-months. Therapists will be either a registered clinical psychologist or a graduate student in clinical psychology under the supervision of a registered clinical psychologist. All treatment will be delivered virtually in the participant's home using the online platform Zoom which is PHIPA/PIPEDA compliant. If participants do not have the technology required for virtual sessions then a tablet will be loaned to them for the duration of treatment. This treatment will be delivered in addition to usual care and no changes to usual care will be required.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria is anyone who meets the criteria of schizophrenia, schizoaffective disorder or any other psychotic disorder, are also 18-65 years of age, know how to use a computer, are not abusing drugs or alcohol and can read and speak English. Participants must be experiencing active symptoms of psychosis as indicated on the PANSS.

Exclusion Criteria:

Exclusion criteria include anyone who has received CBT in the past 6 months, or anyone with a neurological disease or neurological damage that would make it difficult to participate in a talk therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) Total Score | Change from Baseline to Follow-up (6 months post treatment)
  The PANSS is a 30-item semi-structured interview assessing positive, negative symptoms and general psychopathology. Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate severe, 6 = severe, 7 = extreme). The lowest score would be a 30 and the highest score would be 210. A higher score would indicate increased symptomology.

SECONDARY OUTCOMES:
Personal and Social Performance Scale (PSP) | Change from Baseline to Follow-up (6 months post treatment)
  The PSP assesses community functioning through a brief interview with the participant about their daily activities. It contains 4 areas: (1) socially useful activities; including work and study; (2) personal and social relationships; (3) self-care; (4) disturbing and aggressive behaviors. The total score ranges from 1 to 100 and is interpreted on a 10-point intervals. Lower scores indicates more severe functional impairment while higher scores indicate better functioning.
The Psychotic Symptom Rating Scales (PSYRATS) | Change from Baseline to Follow-up (6 months post treatment)
  The PSYRATS assesses frequency and distress associated with the experiences of auditory hallucinations and delusions based on the PANSS interview. Each of the 17 items is scored on a 5-point scale, where a score of 0 indicates no presence, and 4 indicates the highest severity. The lowest score would be a 0 and the highest score would be 68. A higher score would indicate increased symptomology.
Calgary Depression Scale for Schizophrenia (CDSS) | Change from Baseline to Follow-up (6 months post treatment)
  The CDSS is a 9-item interview-based measure of depression symptoms specifically designed for use with people experiencing schizophrenia. Each item is scored on a 4-point scale (0 = absent, 1 = mild, 2 = moderate, 4 = severe). The lowest score would be a 0 and the highest score would be 36. A higher score would indicate increased severity of depressive symptoms.
The Questionnaire About the Process of Recovery (QPR) | Change from Baseline to Follow-up (6 months post treatment)
  The QPR is a self-report measure assessing recovery with people experiencing psychosis. This version contains 22 items while the response to each statement is scored on a 5-point Likert scale ranging from "0 = strongly disagree" to "4 = strongly agree". The lowest possible score is 0 and the highest score could be 88. Higher scores would indicate better recovery.
Beliefs About Paranoia Scale (BAPS) | Change from Baseline to Follow-up (6 months post treatment)
  The BAPS is a 31-item self-report measure assessing metacognitive beliefs about paranoia. The degree of agreement to each statement is scored on a 4-point scale (1 = not at all, 2 = somewhat, 3 = moderately so, 4 = very much). Scales include positive, negative and normalizing beliefs about paranoia, and paranoia as a survival strategy. The lowest score would be 31 and the highest score would be 124. Higher scores are indicative of more beliefs and are shown to be related to paranoid ideation.
Beliefs About Voices Questionnaire (BAVQ) | Change from Baseline to Follow-up (6 months post treatment)
  The BAVQ-R is a 35-item self-report measure assessing metacognitive perception, feelings about and reaction to auditory hallucinations. The degree of agreement to each statement is scored on a 4-point scale, ranging from disagree to strongly agree. Five subscales (malevolence, benevolence, omnipotence, resistance, engagement) are included. The lowest possible score is 0 and the highest score would be 105. Higher scores would indicate a tighter relationship with voices.
Experiences Questionnaire (EQ) | Change from Baseline to Follow-up (6 months post treatment)
  The EQ is a 11-item self-report measure assessing decentering which is the process of distancing one's self from their thoughts and is associated with mindfulness. Frequency of experiences is scored on a 5-point scale, ranging from "1 = never" to "5 = all the time". The lowest possible score is 11 while the highest score would be 55. Higher scores would indicate increased levels of self-acceptance and mindfulness.
Brief Core Schema Scale (BCSS) | Change from Baseline to Follow-up (6 months post treatment)
  The BCSS is a 24-item self-report measure assessing positive and negative judgments individuals hold about themselves and others. Responses are first given dichotomously as "no" or "yes". "No" is scored as 0 and if the answers are "yes", the intensity of beliefs are then rated on a 4-point scale (1 = believe it slightly, 2 = believe it moderately, 3 = believe it very much, 4 = believe it totally). The lowest score would be a 0 and the highest score would be a 96. Higher scores in the positive-self subscale indicate more positive beliefs about selves, while higher scores in the negative-self subscale indicate more negative beliefs about selves. Higher scores in the positive-others subscale indicate more positive beliefs about others, while higher scores in the negative-others subscale indicate more negative beliefs about others.
Dysfunctional Attitude Scale (DAS) | Change from Baseline to Follow-up (6 months post treatment)
  The DAS is a 40-item self-report measure assessing dysfunctional beliefs. The degree of agreement to each statement is scored on a 7-point Likert scale (1 = agree totally, 2 = agree very much, 3 = agree slightly, 4 = neutral, 5 = disagree slightly, 6 = disagree very much, 7 = disagree totally). The lowest possible scale is 40 while the highest possible scale is 280. Higher scores would indicate more negative beliefs.
Davos Assessment of Cognitive Biases Scale (DACOBS) | Change from Baseline to Follow-up (6 months post treatment)
  The DACOBS is a 42-item self-report inventory assessing cognitive processing biases associated with psychosis. The degree of agreement to each statement is scored on a 7-point Likert scale, ranging from "1 = strongly disagree" to "7 = strongly agree". The lowest score would be a 42 and the highest score would be a 294. Higher scores would indicate more cognitive biases.
Childhood Trauma Questionnaire (CTQ) | Change from Baseline to Follow-up (6 months post treatment)
  The CTQ is a 28-item self-report measure assessing experiences of trauma during childhood. Frequency of experiences is reported on a 5-point scale, ranging from "never true" to "very often true". Reverse-coded items are included. The lowest score would be a 28 and the highest score would be a 140. Higher scores would indicate more trauma exposure.
Working Alliance Inventory (WAI) | Change from Baseline to Follow-up (6 months post treatment)
  The WAI assesses the quality of the therapeutic relationship. 36 items are to be completed both by the therapist and the client. Frequency of experiences are rated on a 7-point Likert scale (1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always). Reverse-coded items are included. The lowest score would be a 36 and the highest score would be a 252. Highest scores would indicate more therapeutic alliance.
Psychological Distance Scaling Task (PDST) | Change from Baseline to Follow-up (6 months post treatment)
  The PDST is an experimental task associated with cognitive processing biases in psychosis. It gives measure of both how positive and negative a person views themselves, and how tightly held these beliefs are based on the clustering of the ratings. Participants would place adjectives on the grid based on self-descriptiveness and valence, while responses ranging from "not at all like me" to "very much like me" and "very negative" to "very positive". Smaller interstimulus distances among negative self-relevant adjectives and greater interstimulus distances among positive self-relevant adjectives would indicate more negative biases about selves.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Best, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto Scarborough, Scarborough Village, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu EQ, Birnbaum HG, Shi L, Ball DE, Kessler RC, Moulis M, Aggarwal J. The economic burden of schizophrenia in the United States in 2002. J Clin Psychiatry. 2005 Sep;66(9):1122-9. doi: 10.4088/jcp.v66n0906. PMID 16187769
- [Background] Palmer BA, Pankratz VS, Bostwick JM. The lifetime risk of suicide in schizophrenia: a reexamination. Arch Gen Psychiatry. 2005 Mar;62(3):247-53. doi: 10.1001/archpsyc.62.3.247. PMID 15753237
- [Background] Eack SM, Newhill CE. Psychiatric symptoms and quality of life in schizophrenia: a meta-analysis. Schizophr Bull. 2007 Sep;33(5):1225-37. doi: 10.1093/schbul/sbl071. Epub 2007 Jan 4. PMID 17204532
- [Background] Swartz MS, Perkins DO, Stroup TS, Davis SM, Capuano G, Rosenheck RA, Reimherr F, McGee MF, Keefe RS, McEvoy JP, Hsiao JK, Lieberman JA; CATIE Investigators. Effects of antipsychotic medications on psychosocial functioning in patients with chronic schizophrenia: findings from the NIMH CATIE study. Am J Psychiatry. 2007 Mar;164(3):428-36. doi: 10.1176/ajp.2007.164.3.428. PMID 17329467
- [Background] Chadwick P. Person-based cognitive therapy for distressing psychosis. (Wiley & Sons Ltd., 2006).
- [Background] Kingdon DG, Turkington D. Cognitive Therapy of Schizophrenia. The Guilford Press, 2005.
- [Background] Morrison AP, Renton JC, Dunn H, Williams S, Bentall RP. Cognitive Therapy for Psychosis: A Formulation-Based Approach. Routledge, 2004
- [Background] van der Gaag M, Valmaggia LR, Smit F. The effects of individually tailored formulation-based cognitive behavioural therapy in auditory hallucinations and delusions: a meta-analysis. Schizophr Res. 2014 Jun;156(1):30-7. doi: 10.1016/j.schres.2014.03.016. Epub 2014 Apr 14. PMID 24731619
- [Background] Burns AM, Erickson DH, Brenner CA. Cognitive-behavioral therapy for medication-resistant psychosis: a meta-analytic review. Psychiatr Serv. 2014 Jul;65(7):874-80. doi: 10.1176/appi.ps.201300213. PMID 24686725
- [Background] Velthorst E, Koeter M, van der Gaag M, Nieman DH, Fett AK, Smit F, Staring AB, Meijer C, de Haan L. Adapted cognitive-behavioural therapy required for targeting negative symptoms in schizophrenia: meta-analysis and meta-regression. Psychol Med. 2015 Feb;45(3):453-65. doi: 10.1017/S0033291714001147. Epub 2014 May 22. PMID 24993642
- [Background] Psychosis and schizophrenia in adults: prevention and management. London: National Institute for Health and Care Excellence (NICE); 2014 Mar. Available from http://www.ncbi.nlm.nih.gov/books/NBK555203/ PMID 32207892
- [Background] Norman R, Lecomte T, Addington D, Anderson E. Canadian Treatment Guidelines on Psychosocial Treatment of Schizophrenia in Adults. Can J Psychiatry. 2017 Sep;62(9):617-623. doi: 10.1177/0706743717719894. Epub 2017 Jul 13. PMID 28703017
- [Background] Grant PM, Huh GA, Perivoliotis D, Stolar NM, Beck AT. Randomized trial to evaluate the efficacy of cognitive therapy for low-functioning patients with schizophrenia. Arch Gen Psychiatry. 2012 Feb;69(2):121-7. doi: 10.1001/archgenpsychiatry.2011.129. Epub 2011 Oct 3. PMID 21969420
- [Background] Morrison AP, Law H, Carter L, Sellers R, Emsley R, Pyle M, French P, Shiers D, Yung AR, Murphy EK, Holden N, Steele A, Bowe SE, Palmier-Claus J, Brooks V, Byrne R, Davies L, Haddad PM. Antipsychotic drugs versus cognitive behavioural therapy versus a combination of both in people with psychosis: a randomised controlled pilot and feasibility study. Lancet Psychiatry. 2018 May;5(5):411-423. doi: 10.1016/S2215-0366(18)30096-8. Epub 2018 Apr 5. PMID 29605187
- [Background] Best MW, CIHR Knowledge Synthesis: Examining the Efficacy of Psychosocial Interventions for Schizophrenia-Spectrum disorders delivered through virtual care. 2020.
- [Background] Morrison AP, Renton JC, Dunn H, Williams S, Bentall RP. Cognitive therapy for psychosis: A formulation-based approach. Routledge, 2004.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Nasrallah H, Morosini P, Gagnon DD. Reliability, validity and ability to detect change of the Personal and Social Performance scale in patients with stable schizophrenia. Psychiatry Res. 2008 Nov 30;161(2):213-24. doi: 10.1016/j.psychres.2007.11.012. Epub 2008 Oct 11. PMID 18848731
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Beck AT, Weissman F. Dysfunctional Attitudes Scale (DAS). 1987.
- [Background] van der Gaag M, Schutz C, Ten Napel A, Landa Y, Delespaul P, Bak M, Tschacher W, de Hert M. Development of the Davos assessment of cognitive biases scale (DACOBS). Schizophr Res. 2013 Mar;144(1-3):63-71. doi: 10.1016/j.schres.2012.12.010. Epub 2013 Jan 15. PMID 23332365
- [Background] Bernstein DP, Fink L, Handelsman L, Foote J. Childhood trauma questionnaire. Assessment of family violence: A handbook for researchers and practitioners. 1998.
- [Background] Horvath AO, Greenberg LS. Development and validation of the Working Alliance Inventory. Journal of Counselling Psychology. 1989; 36(2): 223.
- [Background] Ross RM, McKay R, Coltheart M, Langdon R. Jumping to Conclusions About the Beads Task? A Meta-analysis of Delusional Ideation and Data-Gathering. Schizophr Bull. 2015 Sep;41(5):1183-91. doi: 10.1093/schbul/sbu187. Epub 2015 Jan 22. PMID 25616503
- [Background] Diehl C, Yin S, Markell H, Gallop R, Gibbons MBC, Crits-Christoph P. The Measurement of Cognitive Schemas: Validation of the Psychological Distance Scaling Task in a Community Mental Health Sample. Int J Cogn Ther. 2017;10(1):17-33. doi: 10.1521/ijct_2016_09_18. PMID 29250215
- [Background] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819
- [Background] Best MW, Gale D, Tran T, Haque MK, Bowie CR. Brief executive function training for individuals with severe mental illness: Effects on EEG synchronization and executive functioning. Schizophr Res. 2019 Jan;203:32-40. doi: 10.1016/j.schres.2017.08.052. Epub 2017 Sep 19. PMID 28931460